CLINICAL TRIAL: NCT04128553
Title: The Effect of Nurse-led Motivational Interviewing Based on the Trans-theoretical Model on Promoting Physical Activity in Healthy Older Adults: A Randomised Controlled Trial
Brief Title: The Effect of Nurse-led Motivational Interviewing Based on the Trans-theoretical Model
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Gazi University (Other)
Responsible Party: Principal Investigator, Ebru SÖNMEZ, Principal Investigator, Gazi University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: ESONMEZ
Record Dates: First submitted 2019-10-11; First posted 2019-10-16 (Actual); Last update posted 2022-08-01 (Actual); Status verified 2022-07

CONDITIONS: Older Adult; Motivational Interviewing; Physical Activity; Nursing Caries
Keywords: older adult; motivational interviewing; Transtheoretical model; physical activity; nursing
MeSH Terms: conditions — Motor Activity

STUDY DESIGN:
Who Masked: Outcomes Assessor
Masking Description: No researcher and participant blindness were performed.
  The data were collected and recorded by an independent researcher who was trained by the researcher and did not know the groups. The statistics were performed by an independent statistician.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention motivational interview group (Experimental): Face-to-face motivational interviews lasted for an average of 30 minutes. After the MI, the exercise information guideline prepared by the researcher and the TTM-based MI guideline according to the stages were given to the older adults. During the MI, a form prepared by the researcher was used to note the content of the interview. At the end of MI, the next appointment was planned. In addition, the older adults were given a chart prepared by the researcher to note their walk.
  On the other hand, the phone-based motivation interviews lasted an average of five to seven minutes. Before the telephone interview, it was determined which stage of change the older adult was in. Then a motivational interview was held according to the stage.
  Interventions: Behavioral: Intervention motivational interview group
- Control (No Intervention): The Control Group (CG) was only followed up at the beginning and end of the study, no intervention was made. The CG received standard care. Although the family health staff do not give routine and standard training about the benefits of exercising in the FHC to the elderly, they give information when necessary.

INTERVENTIONS:
Behavioral: Intervention motivational interview group — Motivational interviewing (MI) a client-centered, goal-oriented method for enhancing intrinsic motivation to change by exploring and resolving ambivalence. Motivational interviewing is underpinned by a series of principles that emphasise a collaborative therapeutic relationship in which the autonomy of the patient is respected and the patient's intrinsic resources for change are elicited by the therapist.
  In the present study, an effort was made to help the IG to realize the dilemmas of individuals in the precontemplation stage about exercising, and individuals in the contemplation stage to produce their own solutions. In this direction, techniques such as decision balance, importance, and trust technique were applied, thus enabling them to reveal their feelings, thoughts, and reactions regarding the benefits/harms of doing/not doing exercise. They were supported to raise awareness about the consequences and solutions of the causes.
  Arms: Intervention motivational interview group

SUMMARY:
Older adults constitute the age group that leads the most sedentary life in society and is mostly affected by physical inactivity.

This study was conducted to determine how nurse-led Motivational Interviewing (MI) based on the Trans-Theoretical Model (TTM) affected promoting physical activity in older adults.

A randomised controlled trial. The population of this trial was composed of seniors aged between 65 and74 living in a family health center area in Yozgat, Turkey (N=1630). The study sample, estimated via power analysis (d=0.30; 1-β=0.80; α=0.05), constituted 117 older adults (Intervention Group (IG) n=58; Control Group (CG) n=59) who met the inclusion criteria. The data were gathered via a questionnaire, TTM-Scales, Physical Activity Scale for Elderly (PASE), KATZ-ADL by an independent researcher who was blinded to the study groups. A pedometer (JP-600) for each senior was used to calculate the average weekly step counts. The data were analyzed via IBM-SPSS version 23.0. Descriptive statistics, student's t-test, paired-samples t-test, Mann Whitney-U, the Wilcoxon Sign, Friedman, Pearson chi-square, and Fisher-Freeman-Halton exact tests were used to analyze the data. Cohen's d and dz formulas were used to calculate the effect sizes.

MI sessions were held every two weeks in IG. No intervention was applied in CG. Significant progress was found in the change stages of IG compared to CG. The mean of step counts was significant in favour of IG, and the effect size was d=0.641. PASE total score increased significantly in IG, and the effect size was dz=0.202.

This trial indicated that after the TTM-based MI, the change stages of the older adults improved, and their exercising behaviours promoted. In conclusion, TTM and MI are recommended to be used by the nurses toimprove healthy lifestyle behaviours in older adults, and studies to increase physical activity levels in this population should be conducted for a longer period, and studies with larger sample groups are recommended.

DETAILED DESCRIPTION:
This randomised controlled study was carried out in a Family Health Centre (FHC) region in Turkey between April and November 2019.

The population of the study consisted of older adults aged 65 to 74 years residing in the related FHC region (n=1630). First, their records were examined, and those (n=881), who were determined to meet the inclusion criteria [19] based on these records, were called up and invited to the FHC. The sample size was calculated to be at least 90 individuals (d=0.30; 1-β=0.80; α=0.05). Considering the possibility of the participants' withdrawal from the study, all 117 older adults, who met the inclusion criteria in the population and agreed to participate, were included in the study (Intervention Group n=58; Control Group n=59). Figure 1 shows the Consort Flow Diagram of the study.

After stratifying according to age (65-69, 70-74), gender, and stage of exercise change (contemplation and pre-contemplation stage), the stratified simple randomisation procedure was used. No researcher and participant blindness were performed. The randomisation procedure was conducted via the R programming language version 3.5 (https://cran.r-project.org ) by an independent statistician to prevent selection bias. The data were collected and recorded by an independent researcher who was trained by the researcher and did not know the groups. The statistics were performed by an independent statistician.

The data were collected using the personal information form, the TTM scales (the Exercise Stages of Change Scale, the Exercise Processes of Change Scale, the Decisional BalanceScale for Exercise, and the Exercise Self-efficacy Scale), the PASE, the KATZ Activities of Daily Living (ADL) Scale, and a pedometer.

TTM-based MI and Information Guidelines for Gaining Exercise Behaviour were prepared by the researcher within the scope of the relevant literature.

The guideline was used after consulting five experts in the field of nursing who have research on TTM.

A preliminary application was conducted between September 2018 and January 2019. Filling the forms took about 30 minutes. Preliminary motivational interviews were conducted by the researcher and were recorded. Two experts supervised the records and gave feedback. The individuals who participated in the preliminary session were not included in the study.

An independent research assistant trained by the researcher collected the data in the FHC via the face-to-face interview method, and the researcher conducted motivational interviews (face-to-face and on the phone) between April and November 2019.

In the present study, an effort was made to help the IG to realize the dilemmas of individuals in the precontemplation stage about exercising, and individuals in the contemplation stage to produce their own solutions. In this direction, techniques such as decision balance, importance, and trust technique were applied, thus enabling them to reveal their feelings, thoughts, and reactions regarding the benefits/harms of doing/not doing exercise. They were supported to raise awareness about the consequences and solutions of the causes.

Face-to-face motivational interviews lasted for an average of 30 minutes. After the MI, the exercise information guideline prepared by the researcher and the TTM-based MI guideline according to the stages were given to the older adults. During the MI, a form prepared by the researcher was used to note the content of the interview. At the end of MI, the next appointment was planned. In addition, the older adults were given a chart prepared by the researcher to note their walk.

On the other hand, the phone-based motivation interviews lasted an average of five to seven minutes. Before the telephone interview, it was determined which stage of change the older adult was in. Then a motivational interview was held according to the stage.

The CG was only followed up at the beginning and end of the study, no intervention was made. The CG received standard care. Although the family health staff do not give routine and standard training about the benefits of exercising in the FHC to the elderly, they give information when necessary.

ELIGIBILITY:
Inclusion Criteria:

* 65-74 aged seniors, who will voluntarily participate in the study
* Seniors, at least literate or elementary school graduated
* Seniors, at the pre-contemplation or contemplation stages of exercise behavior change
* No cognitive impairment which affects the interpersonal communication
* No muscle-joint problems to be a barrier for the physical activity
* No neuropsychiatric disorder

Exclusion Criteria:

* Individuals whose age are less than 65 and bigger than 75.
* Seniors whose Mini Mental State Test (MMT) scores under 24 points (Mild Cognitive Impairment)
* Seniors whose Geriatric Depression Scale (GDS) scores above 5 points
* Seniors diagnosed with Cancer, Insulin-dependent Type-2 Diabetes Mellitus, Uncontrolled-Hypertension, Heart Failure, Chronic Obstructive Pulmonary Disease (COPD) and Asthma

Termination Criteria:

• Termination criteria are changing in the mental status of the senior during the follow-ups, requesting for leaving the research at any stage and any situation that requires hospitalization needs of the senior.

Ages: 65 Years to 74 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Older Adult
Enrollment: 117 (Actual)
Dates: Start 2019-04-20 (Actual); Primary Completion 2019-11-20 (Actual); Study Completion 2019-11-20 (Actual)

PRIMARY OUTCOMES:
Measurement of stages of change | Twenty-five weeks
  The transtheoretical model construes change as a process involving progress through a series of five stages.
  Precontemplation is the stage in which people are not intending to take action in the foreseeable future, usually measured as the next 6 months. Contemplation is the stage in which people are intending to change in the next 6 months. Preparation is the stage in which people are intending to take action in the immediate future, usually measured as the next month. Action is the stage in which people have made specific overt modifications in their life styles within the past 6 months. Maintenance is the stage in which people are working to prevent relapse but they do not apply change processes as frequently as do people in action.
  It is expected that there will be progress in the levels of stages of change exercise behaviors of the elderly who have been conducted motivational interviews based on transtheoretical model.

SECONDARY OUTCOMES:
Assessment of physical activity level-Physical Activity Scale for the Elderly | Twenty-five weeks
  Physical Activity Scale for the Elderly was developed for the purpose of evaluating the components of physical activities involving leisure time, work-related activities, and the household.
  Physical Activity Scale for the Elderly is a self-reported questionnaire that consists of 12 questions regarding the frequency and duration of leisure time activity, household activity, and work-related activity during the previous 7-day period. The questions are scored differently. The total Physical Activity Scale for the Elderly score is computed by multiplying either the time spent in each activity (hours per week) or participation (i.e. yes or no) in an activity by empirically derived item weights and then summing the overall activities. The overall Physical Activity Scale for the Elderly score ranges from 0 to 400 or more and high scores show better physical activity levels
  With motivational interviews, an increase is expected in Physical Activity Scale for the Elderly scores.
Assessment of physical activity level-Pedometer monitoring | Twenty-five weeks
  Physical activity levels has been determined through Pedometer monitoring. With motivational interviews, an increase is expected the average number of weekly steps taken with a pedometer (JP-600).

CONTACTS AND LOCATIONS:
Overall Officials: Yeter KİTİŞ, Prof., Study Director — Gazi University
Locations (1):
- Gazi University, Ankara, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No
It has not yet been decided with the responsible investigator whether the IPD will be shared.